CLINICAL TRIAL: NCT02850822
Title: Effect of Chemotherapy vs No Chemotherapy Pre-transplantation for Patients With RAEB-1, RAEB-2 and AML Secondary to MDS (Bone Marrow Blast Cells Less Than 50%) Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Effect of Chemotherapy vs No Chemotherapy Pre-transplant to MDS Undergoing Allo-HSCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Fujian Medical University Union Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Zhujiang Hospital (Other); Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Other Study IDs: Therapy vs Notherapy-MDS-2016
Record Dates: First submitted 2016-07-20; First posted 2016-08-01 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2016-07

CONDITIONS: Myelodysplastic Syndrome; Chemotherapy
Keywords: chemotherapy
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Therapy pre-transplantation: Chemotherapy regimen and/or demethylation drugs(such as decitabine) were given pre-transplantation for patients with RAEB-1, REAB-2 and AML Secondary to MDS (bone marrow blast cells less than 50%).
  Interventions: Drug: Demethylation drug; Drug: Chemotherapy regimen
- No Therapy pre-transplantation: No therapy (chemotherapy or demethylation drugs) was given pre-transplantation for patients with RAEB-1, REAB-2 and AML Secondary to MDS (bone marrow blast cells less than 50%).

INTERVENTIONS:
Drug: Demethylation drug — Demethylation drug,such as Decitabine
  Groups: Therapy pre-transplantation
Drug: Chemotherapy regimen — Chemotherapy regimen,such as CAG, G-CSF 5-10ug/kg/day on days 4 and 17；Aclacinomycin 7mg/m2/day on days 4 and 11；Cytarabine 20mg/m2/day on days 4 and 17.
  Groups: Therapy pre-transplantation

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) appears to be an efficient tool to cure refractory anemia with excess blasts-1 (RAEB-1), refractory anemia with excess blasts-2 (RAEB-2) and acute myeloid leukemia (AML) secondary to myelodysplastic syndrome (MDS). At present, the necessity of chemotherapy pre-transplantation for RAEB-1, RAEB-2 and AML secondary to MDS (bone marrow blast cells less than 50%) undergoing allo-HSCT remains in discussion. In this study, the effects of chemotherapy and no chemotherapy pre-transplantation in patients with RAEB-1, REAB-2 and AML secondary to MDS (bone marrow blast cells less than 50%) undergoing allo-HSCT are evaluated.

DETAILED DESCRIPTION:
Allo-HSCT appears to be an efficient tool to cure patients with MDS and AML secondary to MDS. Decitabine and/or chemotherapy pre-transplantation could reduce the blast cells in bone marrow and improve the complete remission rate. However, decitabine and/or chemotherapy had side effects and might increase treatment-related mortality. At present, the necessity of chemotherapy pre-transplantation for RAEB-1, RAEB-2 and AML secondary to MDS (bone marrow blast cells less than 50%) undergoing allo-HSCT remains in discussion. In this study, the effects of chemotherapy and no chemotherapy pre-transplantation in patients with RAEB-1, REAB-2 and AML secondary to MDS (bone marrow blast cells less than 50%) undergoing allo-HSCT are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* RAEB-1, REAB-2 and AML Secondary to MDS (Bone marrow blast cells less than 50%) undergoing allo-HSCT
* 14-65 years

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: RAEB-1, REAB-2 and AML Secondary to MDS (Bone marrow blast cells less than 50%) undergoing allo-HSCT
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 2 year

SECONDARY OUTCOMES:
relapse rate | 2 year
disease-free survival (DFS) | 2 year
transplant-related mortality (TRM) | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Department of Hematology,Nanfang Hospital, Southern Medical University Guangzhou, Guangdong, China, 510515
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Pan D, Zhao W, Jiang Q, Yin C, He H, Liao L, Ye J, Dai M. Wilms' tumor 1 expression combined with genetic mutations for prognostic assessment in MDS. Leuk Lymphoma. 2023 Apr;64(4):856-864. doi: 10.1080/10428194.2023.2185086. Epub 2023 Mar 11. PMID 36905177